CLINICAL TRIAL: NCT07296913
Title: Characterizing the Effects of the X10D Sole on Walking Behavior in Healthy Subjects
Brief Title: Studying the Effects of the X10D Shoe on Walking in Healthy Adults Aged 50 to 65
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Balgrist Campus AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-00477
Record Dates: First submitted 2025-11-27; First posted 2025-12-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: the Immediate and Long-lasting Effects of the X10D Sole on Important Aspects of Walking Function in Healthy Participants; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional shoe (Experimental)
  Interventions: Device: X10D shoe

INTERVENTIONS:
Device: X10D shoe — In this study, we assess the immediate and long-lasting (3-4 weeks) effects of the X10D shoe on a comprehensive battery of biomechanical parameters during various forms of walking. This will be the first study to provide a detailed characterization of the effects of the X10D shoe on diverse walking parameters in healthy individuals aged 50 to 65 years.

SUMMARY:
The aim of this study is to characterize the biomechanical effects of the X10D sole using objective, quantitative measurement methods.

The walking pattern of many people is becoming increasingly passive, and the muscles of the feet and legs are getting weaker. The X10D shoe is an adapted shoe designed to make walking more active and dynamic again.

This study investigates the detailed biomechanical effects of the X10D shoe on the walking pattern of healthy participants. For this purpose, walking with the X10D shoe will be compared with (1) walking in a control shoe with a neutral sole and (2) walking in the participants' everyday sports shoes.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are:

* Healthy subjects aged 50-65 years
* Ability to walk at minimum 30 minutes at a regular pace without assistance or breaks
* Written informed consent as documented by signature (see informed consent form)

Exclusion Criteria:The exclusion criteria are:

* Women who are pregnant or breast feeding
* Current neurological problems affecting walking function and balance
* Current orthopedic problems affecting upper and lower extremity movements
* History of alcohol abuse or the intake of psychotropic drugs
* History of major cardiac condition (e.g., infarction, insufficiency (NYHA II-IV))
* History of major pulmonary condition (e.g., chronic obstructive pulmonary disease (GOLD II-IV))
* Current major depression or psychosis
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia
* Fever of unknown origin

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-10-03 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
CoP path during ankle-foot roll-over movement as measured by pressure plates integrated in the treadmill | up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist Campus AG, Zurich, Canton of Zurich, Switzerland